CLINICAL TRIAL: NCT06265597
Title: The Effect of Healthy Nutrition and Yoga Program Given to Obese Children on Nutritional Behavior, Physical Activity and Anthropometric Measurements
Brief Title: The Effect of Healthy Nutrition and Yoga Program on Obese Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dilara Şahin, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU-SBE-DŞ-01
Record Dates: First submitted 2023-12-18; First posted 2024-02-20 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Obesity, Childhood
Keywords: Anthropometry; Child; Physical Activity; Obesity; Healthy Nutrition; Yoga
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Obesity | interventions — Diet, Healthy

STUDY DESIGN:
Intervention Model Description: There is a control and intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): It includes obese children who are not given a Healthy Nutrition and Yoga Programs.
- İntervention group (Experimental): It includes obese children who are given Healthy Nutrition and Yoga Programs.
  Interventions: Other: Healthy Nutrition and Yoga Program

INTERVENTIONS:
Other: Healthy Nutrition and Yoga Program — * Healthy Nutrition Program
    * At the beginning of the "Healthy Nutrition and Yoga Program" by the researcher give education to families and children in 3 sessions (Importance of Nutrition in School Age, Obesity in School Age, Nutrition Recommendations for Obese Children).
    * Providing individual counseling to children every 2 weeks from the start of the Healthy Nutrition Program, in cooperation with a nutritionist, in line with the basic healthy eating behavior goals.
    * After the 2nd session of the healthy nutrition education and from the beginning of the Yoga Program, in the 2nd, 4th, 6th, 8th and 10th weeks, children are asked to keep a food diary for 2 weekdays and 1 weekend (Thursday-Friday-Saturday) and planning is made according to reaching basic healthy nutrition behavior goals.
  * Yoga Program *Children's yoga is applied to each group twice a week for 12 weeks.
  Arms: İntervention group

SUMMARY:
This study was planned to examine the effects of a healthy nutrition and yoga program given to obese children on nutritional behavior, physical activity and anthropometric measurements.

DETAILED DESCRIPTION:
The prevalence of childhood obesity as a chronic disease is rapidly increasing all over the world, including low- and middle-income countries. Literature highlights that approximately 40.1 million children worldwide are overweight and, at the same time, overweight and obesity are rapidly increasing in almost every country in the world with no signs of slowing down. According to data, it is reported that the prevalence of overweight and obesity among children has increased from 4% to 18% in the last 41 years, and the number of obese school-age children has increased from 11 million to 124 million and has increased more than 10 times. Published reports state that Turkey's childhood obesity risk score is between 70-80%. It is reported that 30% of obese children become obese when they reach adulthood. In this context, identifying and treating individuals with childhood obesity is of great importance. The basic approach in childhood obesity, which is very difficult to treat, is to focus on changeable factors such as daily physical activity and healthy nutrition in an integrated manner. Although it has been proven in the literature that healthy nutrition and physical activity strategies are effective on obesity management, it has been stated that stabilization of this management is difficult. In addition, it is advocated that a holistic approach is required in obesity management to improve long-term results and maintain fitness. Yoga, used in today's obesity, has gained increasing popularity as a mind-body practice. Yoga mind and body movement approaches have the potential to offer a holistic approach to maintaining wellness. Yoga, a lifestyle-based form of physical exercise for health and wellness, emphasizes low physical impact postures (asana), breathwork (pranayama) and meditation (dhyana), regular body stretching, mind-body awareness, and mindful concentration. The literature has reported that yoga could reduce body mass index (BMI) in overweight/obese individuals. Another study reported that regular yoga practice is associated with weight-related health behaviors that may facilitate healthy weight management, such as healthy eating and moderate or vigorous physical activity. It has been concluded in the literature that yoga reduces the BMI values of obese children and that regular yoga practices may make it easier to prevent weight gain. Although the study results show that yoga-based interventions are promising on child obesity well-designed randomized controlled studies on this subject are needed. This study was planned to examine the effects of a healthy nutrition and yoga program given to obese children on nutritional behavior, physical activity and anthropometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* The child's body mass index is at the 85th percentile and above according to age and gender,
* Do not have any chronic disease that may cause obesity (diabetes mellitus, hypothyroidism, etc.).
* No neurodevelopmental delay,
* Those who agree to participate in the study after they and their parents are informed in detail about the study will be included in the study.

Exclusion Criteria:

* Children who fall outside the inclusion criteria will not take part in the research.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Anthropometric Measurements and Child Follow-up Form | "pre-intervention", "12th week immediately after the intervention"
  This form, created by the researchers, includes height, weight, BMI, waist circumference, body composition device anthropometric measurements, and data on nutrition and physical activity.
Family Nutrition and Physical Activity Scale | "pre-intervention", "12th week immediately after the intervention"
  The scale consists of 20 items and is evaluated on a four-point Likert type scale (1=never/almost never, 2=sometimes, 3=often, 4=very often/always).The total score obtained from the scale varies between 20-80. When comparing the total score, high scores indicate less risky family practices and child behaviors for the child's obesity, while low scores indicate high-risk family environment and practices and child behaviors.
Adolescent Identification Form | "pre-intervention"
  The 15-item questionnaire created by the researchers includes sociodemographic data of the child.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Şahin, MSc, Principal Investigator — Erciyes University Health Sciences Institute
Locations (1):
- Karaman Provincial Directorate of National Education, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No